CLINICAL TRIAL: NCT07124884
Title: COLOSOTO: Single-arm Phase II Study Evaluating 5-fluorouracil Plus Panitumumab (Anti-EGFR) and Sotorasib (KRAS G12C Inhibitor) in First-line Treatment of Patients Non-eligible for a Doublet/Triplet Chemotherapy With Advanced Unresectab
Brief Title: 5-fluorouracil Plus Panitumumab (Anti-EGFR) and Sotorasib (KRAS G12C Inhibitor) in First-line Treatment of Patients Non-eligible for a Doublet/Triplet Chemotherapy With Advanced Unresectab
Acronym: COLOSOTO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Northwest Oncology Cooperative Group(GONO) (Unknown); Arbeitsgemeinschaft fur Internistische Onkologie (Other); Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 107-ENGIC01-COLOSOTO; 2024-514030-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Carcinoma; KRAS G12C Mutation; Unresectable Colorectal Cancer
Keywords: sotorasib; colorectal cancer; KRAS G12C
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5-fluorouracil plus Panitumumab and Sotorasib (Experimental): Each patient receives one treatment cycle every two weeks until disease progression or unacceptable toxicity. Panitumumab is administered at a dose of 6 mg/kg via intravenous infusion over one hour during the first cycle, and over 30 minutes from the second cycle onward. The LV5FU2 regimen includes folinic acid (400 mg/m², or 200 mg/m² if levo-leucovorin is used) as a two-hour IV infusion, followed by a 5-FU bolus (400 mg/m² over 10 minutes), and a continuous 5-FU infusion (2400 mg/m² over 46 hours). Sotorasib is given orally at a dose of 960 mg once daily on a continuous basis.
  Interventions: Drug: Administration of experimental treatment association (sotorasib, panitumumab 5FU)

INTERVENTIONS:
Drug: Administration of experimental treatment association (sotorasib, panitumumab 5FU) — Panitumumab is administered at a dose of 6 mg/kg via intravenous infusion over one hour during the first cycle, and over 30 minutes from the second cycle onward. The LV5FU2 regimen includes folinic acid (400 mg/m², or 200 mg/m² if levo-leucovorin is used) as a two-hour IV infusion, followed by a 5-FU bolus (400 mg/m² over 10 minutes), and a continuous 5-FU infusion (2400 mg/m² over 46 hours). Sotorasib is given orally at a dose of 960 mg once daily on a continuous basis.

SUMMARY:
5-fluorouracil (5-FU) is a standard of care in frail/elderly patients with an unresectable colorectal adenocarcinoma (CRC) in first-line setting. Panitumumab plus Sotorasib are promising in advanced line in KRAS G12C mutated CRC. In this study, We assess the safety and efficacy of 5FU combination with Panitumumab and Sotorasib as first-line treatment in frail/elderly patients with unresectable KRAS G12C mutated CRC

DETAILED DESCRIPTION:
COLOSOTO is a multicenter, open-label, prospective single-arm phase II trial, sponsored and cordinated by the Fédération Francophone de Cancérologie Digestive (FFCD) in collaboration with the ENGIC group (European Network in GastroIntestinal Cancer), evaluating 5-FU plus Panitumumab and Sotorasib as first line treatment in patients with MSS/pMMR KRAS G12C mutated unresectable CRC. Inclusion will begin in September 2025, for 36 months. Overall, patients from 40 European sites will be included (in France, Germany, Italy and Spain).

The main inclusion and exclusion criteria are summarized in Table 1. Main inclusion criteria are patients ≥18 years old, with unresectable MSS/pMMR KRASG12C metastatic CRC histologically proven, with altered WHO Performance Status...

Eligible patients will receive LV5FU2 (a 400mg/m2 intravenous (IV) bolus of 5-FU at day 1 (D1) with 400mg/m2 of folinic acid, followed by a continuous 5-FU infusion of 2400mg/m2 over 46 hours) plus Panitumumab (6mg/kg IV at D1) and Sotorasib (960mg PO once daily, every day) in 2-week-cycles (Q2W) until progression or intolerance (cf Figure 1).

Adverse events requiring dose adjustment or treatment discontinuation will all be assessed using the NCI-CTCAE v5.0 scale and manage in accordance with the standard guidelines and the "Summaries of Product Characteristics".

The primary objective is to evaluate the progression-free survival (PFS) of 5FU plus Panitumumab and Sotorasib at 8 months in first-line treatment of patients non-eligible for a doublet/triplet chemotherapy with advanced unresectable KRAS G12C mutated CRC. The progression will be defined as the radiological progression according to RECIST v1.1 criteria assessed by the investigator. A centralized review of CT-scans will be performed to confirm RECIST 1.1 criteria.

Secondary objectives include median progression-free survival (mPFS), disease control rate (DCR), time to progression (TTP), overall survival (OS), best objective response rate (ORR), duration of response (DoR), safety profile, Quality of life (QoL) (with EORTC QLQC30 and FACIT-GP5 questionnaires), and Geriatric assessment (based on G8 score and " Geriatric COre Data sEt " (G-CODE)).

Toxicity will all be evaluated according to the National cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.0) scale. A safety analysis will be done when 10 patients have been treated for at least 2 months to check the good tolerability of 5-FU plus Panitumumab and Sotorasib combination

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically proven advanced-stage unresectable locally advanced or metastatic colorectal adenocarcinoma.
* Proven KRAS G12C mutation as locally assessed by means of an IVDR-compliant test
* Agreement to participate to biological studies (blood samples for ctDNA and send tumour block).
* Patient with one these criteria:

Patient with WHO PS=2 Patient between 70 and 75 years old with WHO PS 1 Patient ≥ 75 years old

* Measurable lesion according to the Response Evaluation Criteria in Solid Tumours 1.1 (RECIST 1.1).
* No prior treatment for the metastatic disease. Prior adjuvant chemotherapy is allowed if there is more than 6 months between the end of adjuvant treatment and relapse.
* Adequate organ function: Hemoglobin > 9 g/dl, Absolute neutrophil count > 1500 /mm3, Platelets > 80 000/mm3, Creatinine clearance rate ≥50 mL/min as calculated using MDRD formula, ALT/AST ≤5×ULN and total bilirubin ≤1.5×ULN.
* Ability to understand and sign written informed consent to participate in the study.
* Provides written informed consent for the study.
* Life expectancy >6 months.
* Women of childbearing potential must agree to use contraception during the trial treatment and for at least 6 months after discontinuation of the experimental treatments. Men who have sexual relationship with women of childbearing potential must agree to use contraception during treatment and for at least 3 months after discontinuation of the experimental treatments.
* Patient affiliated to a social security scheme for France, or equivalent for other countries.

Exclusion Criteria:

- Patient with one of these criteria: Patient fit for doublet/triplet regimen Patient with WHO PS 3 or 4 Patient < 75 years old with WHO PS 0 Patient < 70 years old with WHO PS 0 or 1

* Uncontrolled intercurrent illness including liver (liver cirrhosis Child Pugh B or C) and lung (one second forced expiratory volume <50%) severe insufficiency.
* Patients with high microsatellite instability (MSI-H) or a tumour with mismatched repair (dMMR).
* Clinically significant cardiac abnormalities including prior history of any of the following: severe cardiomyopathy, congestive heart failure of New York Heart Association grade ≥3, history of clinically significant (i.e., active) atherosclerotic cardiovascular disease (myocardial infarction, unstable angina, cerebrovascular accident within 6 months prior to the first dose of study treatments).
* Patients with Dihydropyrimidine Dehydrogenase (DPD) enzyme deficiencies (uracilemia ≥ 16 ng/mL).
* Immunotherapy within 3 months before the beginning of the treatment study.
* Patient under treatment by strong CYP3A4 inducers.
* Patients treated by brivudine within 4 weeks before the first dose of study treatment, or concomitant treatment with brivudine.
* Patient with potentially serious infection.
* Administration of live or live attenuated vaccine within 30 days prior to the first dose of study treatment start.
* Poor nutritional state (albuminemia < 25 g/L or weight loss > 10% during the last month).
* Hereditary problems of galactose intolerance, total lactase deficiency or glucose galactose malabsorption.
* Other malignancy within 2 years prior to study enrolment, except for localized cancer in situ, basal or squamous cell skin cancer adequately treated.
* Less than 4 weeks from major surgeries and not recovered adequately from the procedure and/or any complications from the surgery.
* Patients with persistent toxicities related to prior treatment of grade greater than 1.Is c urrently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks or 5 half-lives (whichever longer) before study entry.
* Hypersensitivity to one of the active substances or to one of the excipients of the trial treatments.
* Patient with interstitial lung disease or pulmonary fibrosis.
* Patients with history of interstitial pneumonitis or pulmonary fibrosis.
* Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study.
* Patient who is under judicial protection and patient who is legally institutionalized or under guardianship or not able to give consent.
* Pregnant or breastfeeding woman.
* Inability to undergo the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patient alive or without progression 8 months after inclusion. | at 8 months after the inclusion.
  Progression will be assessed by the investigator according to recist 1.1 based on images performed every 8 weeks even in case of deferred treatments.
  Clinical progression will not be considered as an event.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years after inclusion.
  Overall survival was defined as the time from the date of inclusion to the patient's death (all causes). For alive patients, the date of the latest news was taken into account.

CONTACTS AND LOCATIONS:
Locations (80):
- France (50):
  - ICO site Paul Papin, Angers
  - Centre Hospitalier Annecy Genevois, Annecy
  - Hôpital Privé, Antony
  - Centre Hospitalier, Aurillac
  - Centre Hospitalier, Bayeux
  - Ch Cote Basque, Bayonne
  - Ch Simone Veille, Beauvais
  - Chu Jean Minjoz, Besançon
  - Polyclinique Courlancy, Bezannes
  - Centre Hospitalier Béthune Beuvry, Béthune
  - Bordeaux Nord Aquitaine, Bordeaux
  - TIVOLI, Bordeaux
  - Chu Morvan, Brest
  - CHU Côte de Nacre, Caen
  - Centre Hospitalier, Cholet
  - Hôpitaux civils, Colmar
  - Polyclinique Saint-Côme, Compiègne
  - Chu Francois Mitterand, Dijon
  - Gf Leclerc, Dijon
  - Institut de cancérologie de Bourgogne GRReCC, Dijon
  - Groupe Hospitalier Mutualiste, Grenoble
  - Chd Vendee, La Roche-sur-Yon
  - Hôpital Franco Britannique, Levallois-Perret
  - Hôpital Privé Le Bois, Lille
  - CHU Dupuytren, Limoges
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Hôpital Jean Mermoz, Lyon
  - Chu La Timone, Marseille
  - Hôpital Européen, Marseille
  - CHRU, Nancy
  - Gh Nord Essone, Orsay
  - Chu Cochin, Paris
  - HEGP, Paris
  - Montsouris, Paris
  - Saint-Louis, Paris
  - Centre Hospitalier, Pau
  - CHU Haut Leveque, Pessac
  - Centre Cario, Plérin
  - Chu La Miletrie, Poitiers
  - CH Quimper Concarneau, Quimper
  - Cac Jean Godinot, Reims
  - Chu Robert Debré, Reims
  - Centre Hospitalier, Saint-Denis
  - Hôpital Privé, Saint-Grégoire
  - Hia Begin, Saint-Mandé
  - Groupe Hospitalier Rance Emeraude, St-Malo
  - Clinique Sainte-Anne, Strasbourg
  - ICANS, Strasbourg
  - CHRU Trousseau, Tours
  - Hôpital Nord Ouest, Villefranche-sur-Saône
- Germany (4):
  - Saint Joseph Hospital Bochum, Bochum
  - Krankenhaus Nordwest-CH Frankfurt Am Main, Frankfurt
  - Universitätsmedizin Göttingen CHU, Göttingen
  - Hämatologisch Onkologische Praxis Eppendorf, Hamburg
- Italy (17):
  - Centro Di Riferimento Oncologico Di Aviano, Aviano
  - Azienda Ospedaliero Universitaria Policlinico Rodolico San Marco Di Catania, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Unita Sanitaria Locale 6 Livorno, Livorno
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan
  - Azienda Ospedaliero-Universitatia Di Cagliari, Monserrato
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda USL Toscana Centro, Prato
  - Azienda Unita Sanitaria Locale Della Romagna, Ravenna
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero-Universitaria Città della salute e della scienza di Torino Presidio Molinette, Torino
  - Pia Fondazione Di Culto E Religione Card Panico, Tricase
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Instituto Catalan de Oncologia. Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Clinico San Carlos, San Carlos
  - Consorcio Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No